CLINICAL TRIAL: NCT05675917
Title: Feasibility and Acceptability of the MacuTest Website for Personalized AMD Risk Prediction and Prevention: Pilot Study
Brief Title: MacuTest Website for Personalized AMD Risk Prediction and Prevention
Acronym: MACUTEST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative issues
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/46
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Macular Degeneration
Keywords: Macular degeneration; prediction; digital platform; personalized medicine
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MacuTest website (Experimental): The MacuTest platform will be used to collect the data needed to predict AMD risk. AMD risk prediction is evaluated by a mathematical algorithm based on the data collected and integrated into the platform.
  The ophthalmologist will fill in the ophthalmologist questionnaire in the platform with data on the fundus and blood pressure, after examining the patient.
  The patient will fill in the lifestyle questionnaires (nutrition, smoking, gender, year of birth, level of education) with his personal equipment (computer, smartphone or tablet).
  Interventions: Device: MacuTest platform

INTERVENTIONS:
Device: MacuTest platform — The MacuTest platform will be used to collect the data needed to predict AMD risk. AMD risk prediction is evaluated by a mathematical algorithm based on the data collected and integrated into the platform.
  The ophthalmologist will fill in the ophthalmologist questionnaire in the platform with data on the fundus and blood pressure, after examining the patient.
  The patient will fill in the lifestyle questionnaires (nutrition, smoking, gender, year of birth, level of education) with his personal equipment (computer, smartphone or tablet).

SUMMARY:
LEHA team of Bordeaux University has developed an Age-related Macular Degeneration (AMD) prediction algorithm (taking into account age, 49 genetic variants, the presence of early retinal abnormalities, tobacco consumption, food quality, blood pressure and education level) and is currently developing the MacuTest website, integrating this prediction algorithm. This platform offers participants the possibility to enter their personal lifestyle data, to couple them with an ophthalmological examination and a genetic test, in order to evaluate their personalized risk of AMD. The main objective of this pilot study is to evaluate the feasibility of estimating the predicted AMD risk

DETAILED DESCRIPTION:
AMD is the leading cause of blindness in industrialized countries. Current treatments only address the neovascular form and do not always prevent vision loss. This multifactorial pathology involves both genetic factors (more than 50 loci identified) and environmental factors. The genes identified suggest an important contribution of inflammation and innate immunity as well as lipid metabolism in the physiopathology of AMD. As a potential target for preventive actions, the role of lifestyle has also been the subject of much work. Thus, epidemiological studies have identified smoking as an important risk factor. The role of nutrition and metabolism in ocular aging is of growing interest, with hypotheses focusing more specifically on the joint effect of antioxidants and lipids. It is therefore important to develop prevention strategies. In this context, it is necessary to be able to identify at an early stage those people most at risk of developing AMD, in order to propose interventions aimed at reducing the risk of visual loss (reinforced ophthalmological follow-up for rapid detection and treatment of neovascular forms, lifestyle recommendations, nutritional supplementation, etc.).

During the baseline (V1) and the 12-months follow-up (V3) visits, lifestyle data (tobacco, diet, education) will be collected within online self-questionnaires on the MacuTest platform. Ophthalmological examination with evaluation of retinal anomalies, blood pressure, and saliva collection (inclusion only) for genetic testing will be perform by the ophthalmologist.

At the 6-months follow-up visit (V2), the ophthalmologist will give the participant the results of the genetic test and explanations and interpretation of the results he or she deems necessary.

At the 12-months follow-up visit (V3), the participant will fill in a questionnaire to evaluate the MacuTest platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older of European geographic origin
* Presence of early signs of AMD (drusen and/or pigment abnormalities) and/or parents with advanced AMD.
* Absence of any advanced form of AMD (atrophic or neovascular AMD).
* Patient who can read, understand and speak French.
* Patient with access to the MacuTest internet platform throughout the study (telephone, tablet, computer).
* Patient with the ability and willingness to carry out all planned visits and assessments.
* Patient with health insurance.
* Signed informed consent.

Exclusion Criteria:

* Presence of a severe ocular pathology that prevents an examination of the fundus.
* Patient with a history of a medical condition that, in the opinion of the investigator, would prevent the completion of scheduled study visits and completion of the study.
* Adult under legal protection or residing in a health or social institution.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
estimation of AMD risk | Month 6
  Percentage of participants who received an estimation of their risk of AMD

SECONDARY OUTCOMES:
Socio-demographic characteristics | baseline
  Socio-demographic characteristics (age, gender, education level)
Lifestyle characteristics | baseline
  Lifestyle characteristics (tobacco use, diet quality)
Ophthalmological characteristics | baseline
  Ophthalmological characteristics (presence of drusen, pigmentary abnormalities, advanced AMD in each eye)
Genetic risk | baseline
  Evaluated by the presence or not of the following variants: CFH_rs187328863 ; CFH_rs570618 ; CFH_rs148553336 ; CFH_rs10922109 ; CFH_rs35292876 ; CFH_rs121913059 ; CFH_rs61818925 ; CFH_rs191281603 ; COL4A3_rs11884770 ; ADAMTS9_rs62247658 ; COL8A1_rs140647181 ; COL8A1_rs55975637 ; CFI_rs10033900 ; CFI_rs141853578 ; PRLR_SPEF2_rs114092250 ; C9_rs62358361 ; C2_rs144629244 ; C2_rs429608 ; C2_rs181705462 ; C2_rs114254831 ; C2_rs943080 ; PILRB_rs7803454 ; KMT2E_rs1142 ; TNFRSF10A_rs79037040 ; MIR6130_rs10781182 ; TGFBR1_rs1626340 ; ABCA1_rs2740488 ; ARHGAP21_rs12357257 ; ARMS2_rs3750846 ; RDH5_rs3138141 ; ACAD10_rs61941274 ; B3GALTL_rs9564692 ; RAD51B_rs61985136 ; RAD51B_rs2842339 ; LIPC_rs2043085 ; LIPC_rs2070895 ; CETP_rs17231506 ; CETP_rs5817082 ; CTRB2_rs72802342 ; TMEM97_rs11080055 ; NPLOC4_rs6565597 ; C3_rs12019136 ; C3_rs147859257 ; C3_rs2230199 ; APOE_rs429358 ; APOE_rs73036519 ; C20orf85_rs201459901_ ; SYN3_rs5754227 ; SLC16A8_rs8135665 ;

IPD SHARING:
Plan to Share IPD: No